CLINICAL TRIAL: NCT07117188
Title: Observational Analysis of the Associational Between Dietary Factors and Postprandial Glucose Fluctuations
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: United Imaging Healthcare (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20250519040454800
Record Dates: First submitted 2025-08-04; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- diabetes cohort
- Non-diabetic cohort

SUMMARY:
This study aims to observe the differences in postprandial blood glucose fluctuations in patients with type 2 diabetes and healthy individuals after consuming different dietary recipes through a prospective cohort study, in order to optimize individualized dietary strategies.

ELIGIBILITY:
Inclusion Criteria:

* For diabetes cohort:

  1. diagnosed with type 2 diabetes is more than one month
  2. Glycated hemoglobin (HbA1c) : 6.5%<HbA1c<10.5%(48 mmol/mol < HbA1c < 91.3 mmol/mol)
  3. Requirements for the blood glucose management plan: Within one month before the start of the trial, a simple lifestyle, and/or one or more oral hypoglycemic drugs (metformin, DPP-4 inhibitors, SGLT-2 inhibitors, TZD drugs, GLP-1 receptor agonists), and/or basal insulin treatment once a day were adopted, and the regimen was required to be maintained stably within 7 days before the start of the trial and during the trial.
  4. Take the test voluntarily and sign the informed consent form.
* For Non-diabetic cohort:

  1. Glycated hemoglobin (HbA1c) : HbA1c<5.7%
  2. Fasting blood glucose was between 3.9 and 5.6 mmol/L, and 2-hour postprandial blood glucose was less than 7.8mmol/L
  3. Take the test voluntarily and sign the informed consent form.

Exclusion Criteria:

1. Skin damage, scars, redness and swelling at the wearing site, or those with subcutaneous edema at the wearing site of an infected person, or those allergic to disinfectants, medical adhesive tapes or patches.
2. Epilepsy or cognitive impairment, immunosuppressive disorders, and systemic neurological diseases.
3. Required emergency or inpatient treatment due to severe hypoglycemia (blood glucose < 3.0mmol/L with consciousness disorder), diabetic ketoacidosis, or non-ketotic hyperosmolar syndrome in the past six months.
4. Severe circulatory disorders.
5. Long-term gastrointestinal diseases (such as celiac disease, gastroparesis, etc.), or eating disorders or having undergone bariatric surgery (such as gastric bypass surgery); Has a history of severe infection within the past month; History of malignant tumors (except skin cancer); Mental illnesses such as depression; Severe liver and kidney dysfunction (renal function: estimated eGFR<30mL/min or maintenance dialysis required;) Liver function: ALT and AST>3 times the upper limit of the normal value or active liver disease. History of severe cardiovascular disease (NYHA cardiac function classification III-IV or BNP >400 pg/mL).
6. Technical or language barriers: Inability to use research applications or understand text; Unable to cooperate with the use of research equipment such as continuous blood glucose monitors and accelerometers.
7. Drug use: Immunosuppressants, proton pump inhibitors, or steroid drugs have been used in the past 4 weeks or are planned to be used during the study period.
8. BMI<16.5 kg/m².
9. Magnetic resonance imaging (MRI) examination is planned or conducted within 16 days of product use.
10. Pregnant and lactating women, and those planning to become pregnant during the study period.
11. Those whom the researchers consider unsuitable to participate in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study recruited diabetic and non-diabetic individuals aged 18 to 80 in Shanghai, China. The subjects had fixed or no medication regimens and possessed the ability to use and understand new technologies.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
postprandial glycemic response | 14 days
  postprandial glycemic response (PPGR) : PPGR refers to the dynamic changes in blood sugar levels after eating, reflecting the extent to which food affects blood sugar. PPGR is mainly determined by calculating the area under the Incremental curve (Incremental AUC, iAUC) of blood glucose.

SECONDARY OUTCOMES:
postprandial blood glucose peak | 14 days
  The maximum postprandial blood glucose measured by CGM

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No